CLINICAL TRIAL: NCT02352974
Title: Open Label Pilot Trial in Adults With Recent-onset T1D to Evaluate the Safety, Diabetes Status and Immune Response of GAD-antigen (Diamyd®) Therapy Administered Into Lymph Nodes in Combination With an Oral Vitamin D Regimen
Brief Title: GAD-Alum (Diamyd) Administered Into Lymph Nodes in Combination With Vitamin D in Type 1 Diabetes (DIAGNODE-1)
Acronym: DIAGNODE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnny Ludvigsson (Other Government)
Collaborators: Swedish Child Diabetes Foundation (Other); Ostergotland County Council, Sweden (Other); Diamyd Medical AB (Industry)
Responsible Party: Sponsor-Investigator, Johnny Ludvigsson, MD, PhD, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAGNODE-1
Record Dates: First submitted 2014-12-09; First posted 2015-02-02 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diamyd; Diabetes; Juvenile Diabetes; Diabetes Type 1; Type 1 Diabetes; Autoimmune Diabetes; Insulin Dependent Diabetes; Type 1 Diabetes Mellitus; rhGAD65 (Recombinant Human GAD with molecular mass 65,000); GAD65; GAD-Alum; Diabetes Mellitus; Diabetes mellitus Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Vitamin D
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GAD-Alum+Vitamin D (Experimental): GAD-Alum (Diamyd) injected into Lymph Nodes Dosage and interval: One injection of 4 µg Diamyd will be administered into the lymph nodes at three occasions, with one month intervals
  Vitamin D (Calciferol) in oral solution. Dosage and interval: 2000 IU daily for 120 days
  Interventions: Drug: GAD-Alum; Drug: Vitamin D

INTERVENTIONS:
Drug: GAD-Alum
  Other Names: Diamyd
Drug: Vitamin D
  Other Names: Calciferol

SUMMARY:
The objectives of the main study is to:

* Evaluate the safety of giving GAD-Alum (Glutamic acid decarboxylase) (Diamyd) directly into lymph glands in combination with an oral vitamin D regimen
* Evaluate how the above mentioned treatments influence the immune system and endogenous insulin secretion.

The objective of the sub-study is to:

* Evaluate safety after a fourth injection with 4 μg GAD-Alum direct into an inguinal lymph gland in 3 adult patients from the main study
* Evaluate how the above mentioned treatment influences the immune system and endogenous insulin secretion.

DETAILED DESCRIPTION:
Eligible patients will be treated with 4 µg GAD-Alum into an inguinal lymph gland at three occasions, with one month intervals in combination with Vitamin D (14 000 IU/week) for 4 months, starting 1 month prior to first GAD-Alum injection.

A sub-study will include three adult patients from the main study and evaluate safety after a fourth injection with 4 μg GAD-Alum into an inguinal lymph gland in combination with oral vitamin D intake. The Prolonged Extension Study Period is 12 months and will start 30,5 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given by patients
2. Type 1 diabetes according to the ADA (American Diabetes Association) classification with < 6 months diabetes duration
3. Age 12.00-29.99 years at diagnosis of Type 1 diabetes
4. Fasting C-peptide ≥0.12 nmol/L
5. Pos GADA(Antibodies to GAD with molecular mass 65,000) but < 50 000 random units
6. Females must agree to avoid pregnancy and have a negative urine pregnancy test
7. Patients of childbearing potential must agree to using adequate contraception, until 1 year after the last administration of GAD-Alum.

Exclusion Criteria:

1. Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
2. Continuous treatment with any inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
3. Treatment with any oral or injected anti-diabetic medications other than insulin
4. Treatment with Vitamin D, marketed or not, or unwilling to abstain from such medication during the trial
5. A history of anaemia or significantly abnormal haematology results at screening
6. A history of epilepsy, head trauma or cerebro-vascular accident, or clinical features of continuous motor unit activity in proximal muscles
7. Clinically significant history of acute reaction to vaccines or other drugs in the past
8. Treatment with any vaccine, including influenza vaccine, within 4 months prior to planned first study drug dose or planned treatment with any vaccine up to 4 months after the last injection with study drug.
9. Participation in other clinical trials with a new chemical entity within the previous 3 months
10. Inability or unwillingness to comply with the provisions of this protocol
11. A history of alcohol or drug abuse
12. A significant illness other than diabetes within 2 weeks prior to first dosing
13. Known human immunodeficiency virus (HIV) or hepatitis
14. Females who are lactating or pregnant (the possibility of pregnancy must be excluded by urine βHCG (beta-human chorionic gonadotropin) on-site within 24 hours prior to the GAD-Alum treatment)
15. Males or females not willing to use adequate contraception until 1 year after the last GAD-Alum treatment
16. Presence of associated serious disease or condition, including active skin infections that preclude subcutaneous injection, which in the opinion of the investigator makes the patient non-eligible for the study
17. Deemed by the investigator not being able to follow instructions and/or follow the study protocol

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

REFERENCES:
- [Derived] Casas R, Dietrich F, Barcenilla H, Tavira B, Wahlberg J, Achenbach P, Ludvigsson J. Glutamic Acid Decarboxylase Injection Into Lymph Nodes: Beta Cell Function and Immune Responses in Recent Onset Type 1 Diabetes Patients. Front Immunol. 2020 Oct 9;11:564921. doi: 10.3389/fimmu.2020.564921. eCollection 2020. PMID 33162978
- [Derived] Tavira B, Barcenilla H, Wahlberg J, Achenbach P, Ludvigsson J, Casas R. Intralymphatic Glutamic Acid Decarboxylase-Alum Administration Induced Th2-Like-Specific Immunomodulation in Responder Patients: A Pilot Clinical Trial in Type 1 Diabetes. J Diabetes Res. 2018 May 24;2018:9391845. doi: 10.1155/2018/9391845. eCollection 2018. PMID 30009185

RESULTS

PARTICIPANT FLOW:
Groups:
- GAD-Alum+Vitamin D: GAD(Glutamic acid decarboxylase)-Alum (Diamyd) injected into Lymph Nodes Dosage and interval: One injection of 4 µg Diamyd will be administered into the lymph nodes at three occasions, with one month intervals
  Vitamin D (Calciferol) in oral solution. Dosage and interval: 2000 IU daily for 120 days
  GAD-Alum
  Vitamin D
Period: Main Study
Arm/Group | GAD-Alum+Vitamin D
Started | 12
Completed | 12
Not Completed | 0
Period: Extension
Arm/Group | GAD-Alum+Vitamin D
Started | 3 (Only 3 out of the 12 patients who completed the main study continued in to the extension period.)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GAD-Alum+Vitamin D: GAD-Alum (Diamyd) injected into Lymph Nodes Dosage and interval: One injection of 4 µg Diamyd will be administered into the lymph nodes at three occasions, with one month intervals
  Vitamin D (Calciferol) in oral solution. Dosage and interval: 2000 IU daily for 120 days
  GAD-Alum
  Vitamin D
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 12
Weight [Mean (Standard Deviation); unit: kg] | 64.0 (13.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.1 (3.8)
Type 1 diabetes duration [Mean (Standard Deviation); unit: days] | 65.1 (55.1)
GADA (Antibodies to GAD with molecular mass 65,000) [Mean (Standard Deviation); unit: U/mL^2] | 4067.1 (8491.6)
Weighted C-peptide [Mean (Standard Deviation); unit: nmol/L] | 0.55 (0.19)
90-minute C-peptide [Mean (Standard Deviation); unit: nmol/L] | 0.67 (0.19)
Fasting C-peptide [Mean (Standard Deviation); unit: nmol/L] | 0.27 (0.08)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 67.17 (28.17)
Average insulin dose/kg/24 h [Mean (Standard Deviation); unit: IU] | 0.40 (0.20)
IDAA1c [Mean (Standard Deviation); unit: IU/kg/day] | 9.91 (3.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Injection Site Reactions Month 1
Description: Reactions of the injection site (Erythema, Oedema, Haematoma, Tenderness, Pain, Itching)
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
Participants
  Erythema | 0
  Oedema | 0
  Haematoma | 0
  Tenderness | 1
  Pain | 0
  Itching | 0
  Other | 0

2. Primary Outcome: Number of Subjects With Injection Site Reactions Month 2
Description: Reactions of the injection site (Erythema, Oedema, Haematoma, Tenderness, Pain, Itching)
Time Frame: Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
Participants
  Erythema | 0
  Oedema | 0
  Haematoma | 0
  Tenderness | 1
  Pain | 0
  Itching | 0
  Other | 0

3. Primary Outcome: Number of Subjects With Injection Site Reactions Month 3
Description: Reactions of the injection site (Erythema, Oedema, Haematoma, Tenderness, Pain, Itching)
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
Participants
  Erythema | 0
  Oedema | 0
  Haematoma | 0
  Tenderness | 2
  Pain | 0
  Itching | 0
  Other | 0

4. Primary Outcome: Number of Subjects With Injection Site Reactions Month 32
Description: Reactions of the injection site (Erythema, Oedema, Haematoma, Tenderness, Pain, Itching)
Time Frame: Month 32, extension period
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
Participants
  Erythema | 0
  Oedema | 0
  Haematoma | 0
  Tenderness | 0
  Pain | 0
  Itching | 0
  Other | 0

5. Secondary Outcome: Mean Change in C-peptide AUC (Area Under the Curve) (Mean 120min) Value, Month 15
Description: Change from baseline to month 15 in C-peptide AUC (Area Under the Curve) (mean 120min) value
  AUC (mean 120min) (nmol/L) is the C-peptide AUC during an MMTT (nmol/L*minutes) divided by the duration of the MMTT (minutes) i.e. C-peptide weighted average concentration
Time Frame: Baseline to month 15 at 0, 30, 60, 90, 120 minutes post-dose
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.11 (0.12)

6. Secondary Outcome: Mean Change in C-peptide AUC(Mean 120min) Value, Month 30
Description: Change from baseline to month 30 in C-peptide AUC(mean 120min) value
  AUC (mean 120min) (nmol/L) is the C-peptide AUC during an MMTT (nmol/L*minutes) divided by the duration of the MMTT (minutes) i.e. C-peptide weighted average concentration
Time Frame: Baseline to month 30 at 0, 30, 60, 90, 120 minutes post-dose
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.22 (0.16)

7. Secondary Outcome: Mean Change in C-peptide AUC(Mean 120min) Value, Month 43
Description: Change from baseline to month 43 in C-peptide AUC(mean 120min) value
  AUC (mean 120min) (nmol/L) is the C-peptide AUC during an MMTT (nmol/L*minutes) divided by the duration of the MMTT (minutes) i.e. C-peptide weighted average concentration
Time Frame: Baseline to month 43, extension period at 0, 30, 60, 90, 120 minutes post-dose
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
nmol/L | -0.13 (0.05)

8. Secondary Outcome: Mean Change in C-peptide 90-minute Value, Month 15
Description: Change from baseline to month 15 in C-peptide 90-minute value
Time Frame: Baseline to month 15
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.16 (0.15)

9. Secondary Outcome: Mean Change in C-peptide 90-minute Value, Month 30
Description: Change from baseline to month 30 in C-peptide 90-minute value
Time Frame: Baseline to month 30
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.29 (0.17)

10. Secondary Outcome: Mean Change in C-peptide 90-minute Value, Month 43
Description: Change from baseline to month 43 in C-peptide 90-minute value
Time Frame: Baseline to month 43, extension period
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
nmol/L | -0.16 (0.03)

11. Secondary Outcome: Mean Change in Fasting C-peptide Value, Month 15
Description: Change from baseline to month 15 in fasting C-peptide value
Time Frame: Baseline to month 15
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.03 (0.12)

12. Secondary Outcome: Mean Change in Fasting C-peptide Value, Month 30
Description: Change from baseline to month 30 in fasting C-peptide value
Time Frame: Baseline to month 30
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
nmol/L | -0.10 (0.12)

13. Secondary Outcome: Mean Change in Fasting C-peptide Value, Month 43
Description: Change from baseline to month 43 in fasting C-peptide value
Time Frame: Baseline to month 43, extension period
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
nmol/L | -0.07 (0.04)

14. Secondary Outcome: Mean Change in HbA1c, Month 15
Description: Change from baseline to month 15 in HbA1c
Time Frame: Baseline to month 15
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
mmol/mol | -14.25 (18.91)

15. Secondary Outcome: Mean Change in HbA1c, Month 30
Description: Change from baseline to month 30 in HbA1c
Time Frame: Baseline to month 30
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
mmol/mol | -10.67 (18.67)

16. Secondary Outcome: Mean Change in HbA1c, Month 43
Description: Change from baseline to month 43 in HbA1c
Time Frame: Baseline to month 43, extension period
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
mmol/mol | -30.67 (21.22)

17. Secondary Outcome: External Insulin Dose, Baseline
Description: External insulin dose at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 0.36 (0.13)

18. Secondary Outcome: External Insulin Dose, Month 15
Description: External insulin dose at month 15
Time Frame: Month 15
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 0.34 (0.20)

19. Secondary Outcome: External Insulin Dose, Month 30
Description: External insulin dose at month 30
Time Frame: Month 30
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 0.44 (0.22)

20. Secondary Outcome: External Insulin Dose, Month 43
Description: External insulin dose at month 43
Time Frame: Month 43, extension period
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
IU/kg/day | 0.25 (0.02)

21. Secondary Outcome: Mean IDAA1c Values, Baseline
Description: Insulin dose-adjusted HbA1c (IDAA1c)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 9.00 (1.89)

22. Secondary Outcome: Mean IDAA1c Values, Month 15
Description: Insulin dose-adjusted HbA1c (IDAA1c)
Time Frame: Month 15
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 7.64 (0.99)

23. Secondary Outcome: Mean IDAA1c Values, Month 30
Description: Insulin dose-adjusted HbA1c (IDAA1c)
Time Frame: Month 30
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 12
IU/kg/day | 8.36 (1.28)

24. Secondary Outcome: Mean IDAA1c Values, Month 43
Description: Insulin dose-adjusted HbA1c (IDAA1c)
Time Frame: Month 43, extension period
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | GAD-Alum+Vitamin D
Number analyzed (Participants) | 3
IU/kg/day | 7.11 (0.93)

ADVERSE EVENTS:
Time Frame: During main study period (baseline to month 30) and extension (month 37 and 43)
Arm/Group | GAD-Alum+Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-Alum+Vitamin D (N=12)
Retinopathy (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (3)
Pyrexia (General disorders) | 1 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (35)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fascilitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 2 (2)
Panic disorder (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT02352974/Prot_SAP_000.pdf